CLINICAL TRIAL: NCT07184359
Title: The Use of Social Media as an Auxiliary Tool in the Teaching-learning Process of Dental Students
Brief Title: Application of Social Media as a Supporting Tool in the Teaching and Learning Process of Dentistry Students
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Karina Lopes Devito (Other)
Responsible Party: Sponsor-Investigator, Karina Lopes Devito, PhD, Federal University of Juiz de Fora
Organization: Federal University of Juiz de Fora (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CAAE: 74616923.5.0000.5147
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-09

CONDITIONS: Social Media; Dental Education and Teaching Learning Processes
Keywords: Social Media; Dental Education; Radiology; Information and Communication Technology; Teaching Learning Processes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional Learning Group (Active Comparator): Teaching-learning process carried out without the inclusion of supplementary content on social media platforms.
  Interventions: Behavioral: Traditional Learning
- Passive Social Media Supplement Group (Experimental): Teaching-learning process supplemented with content passively accessed through social media.
  Interventions: Behavioral: Traditional Learning; Behavioral: Passive Social Media
- Active Social Media Engagement Group (Experimental): Teaching-learning process supplemented with content actively produced and shared through social media.
  Interventions: Behavioral: Traditional Learning; Behavioral: Passive Social Media; Behavioral: Active Social Media

INTERVENTIONS:
Behavioral: Traditional Learning — All participants will have access to the conventional teaching-learning process (lecture-based classes). These theoretical classes will be delivered as part of the Dental Radiology course. During the semester, the topics covered will include intraoral radiographic techniques, radiographic processing, intraoral radiographic anatomy, and dental and periodontal alterations and lesions.
Behavioral: Passive Social Media — The second group (Passive Social Media Supplement Group) will participate in the conventional teaching-learning process, supplemented by the passive consumption of educational content on social media, produced by the third group. The materials consumed will include the following content: intraoral radiographic techniques, radiographic processing, intraoral radiographic anatomy, and dental and periodontal alterations and lesions.
  Arms: Active Social Media Engagement Group; Passive Social Media Supplement Group
Behavioral: Active Social Media — The third group (Active Social Media Engagement Group) will participate in the conventional teaching-learning process, supplemented by the creation of educational audiovisual materials, which will subsequently be shared on social media and accessed both by their own group and by the second group. The materials will cover the following topics: intraoral radiographic techniques, radiographic processing, intraoral radiographic anatomy, and dental and periodontal alterations and lesions.
  Arms: Active Social Media Engagement Group

SUMMARY:
This study aims to explore dental students' perceptions of the role of Information and Communication Technologies (ICT) in supporting the teaching and learning process, particularly within the university setting. It seeks to identify gaps at the interface between information gathering, education, and ICT, providing valuable insights into students' awareness and acceptance of the content they access. The findings are expected to contribute to optimizing the use of ICT as an educational support tool, strengthening the curriculum, and preparing future dentists to better understand the interaction between ICT and teaching. Ultimately, this will help foster a generation of more qualified professionals.

DETAILED DESCRIPTION:
The sample will consist of 90 undergraduate students from the School of Dentistry at the Federal University of Juiz de Fora (UFJF), aged 18 years or older, who are regularly enrolled in the Dental Radiology course.

Recruitment will take place during the course sessions, through announcements made by the course instructors. The research team will only have access to participants' data after the student voluntarily makes contact and provides their information. All students who express interest and meet the inclusion criteria will be enrolled as volunteers.

Participants will be fully informed about the objectives and procedures of the study and will sign the Informed Consent Form (ICF). Each volunteer will receive a confidential identification number, which will be linked to their responses and will allow the exclusion of their data should they choose to withdraw from the study. Withdrawal may occur at any time, without any harm or disadvantage. In case of withdrawal, the participant need only notify the principal investigator, and their data will be excluded, ensuring the anonymity of all volunteers.

The results will not be presented individually, but only in aggregate form, without any identification of participants. All data collected will be accessible only to the principal investigator and the research team.

After signing the ICF, participants will be randomly allocated, by drawing lots, into three experimental groups:

Traditional Learning Group (n = 30): students undergoing the teaching-learning process without complementary content on social media; Passive Social Media Supplement Group (n = 30): students undergoing the teaching-learning process with complementary content on social media, consumed passively; Active Social Media Engagement Group (n = 30): students undergoing the teaching-learning process with complementary content through the production of audiovisual material, later shared on social media, representing active consumption.

The social media platform used will be the one identified as most frequently accessed by the students in a prior survey. The complementary digital material will cover topics from the Dental Radiology curriculum, including: intraoral radiographic techniques, radiographic processing, intraoral radiographic anatomy, and dental and periodontal alterations and lesions.

The content for G2 will be developed by students from G3, under the supervision of the course instructor and research team member (KLD). For G3, the materials will be produced and posted by the students themselves, after faculty review.

At the end of the activities, students' performance will be assessed through the Objective Structured Clinical Examination (OSCE), composed of five stations simulating clinical situations, with predetermined criteria and timing for each task. The competencies to be assessed will include: a) radiographic techniques; b) dental numbering notation; c) radiographic anatomy; d) radiographic interpretation of caries/restorations; and e) radiographic periodontal diagnosis.

At no stage will individual results be disclosed to other students or to anyone outside the research team. All data will remain restricted to the principal investigator and the research team and will be presented only in aggregate and anonymized form.

ELIGIBILITY:
Inclusion Criteria

* Students aged 18 years or older, of any gender.
* Regular enrollment in the Dental Radiology course at the School of Dentistry, Federal University of Juiz de Fora (UFJF), Juiz de Fora campus.
* Voluntary agreement to participate in the study, confirmed by signing the Informed Consent Form.

Exclusion Criteria

* Students who report audiovisual discomfort when using smartphones or computers.
* Individuals who are not users of social media.
* Lack of internet access.
* Presence of medical or psychological contraindications to the use of electronic devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01-14 (Actual); Primary Completion 2026-01-12 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Overall OSCE Score | The assessment will be conducted at the end of each academic semester, specifically in the 15th week after the beginning of the semester, in accordance with the institution's academic calendar.
  The study will use the Objective Structured Clinical Examination (OSCE) to assess students' clinical competencies in a standardized and objective manner. Participants will rotate through five consecutive stations designed to evaluate specific skills under controlled conditions. One active station will involve performing a periapical radiograph while following biosafety, radioprotection, and processing protocols. Four passive stations will focus on case analysis, interpretation, and clinical decision-making. Each station will include a structured checklist with predefined criteria and will be scored from zero to 100, with 100 being the best result. All participants will complete the stations in the same sequence, and the final score will be calculated by summing the points obtained and dividing by the number of stations, providing a standardized performance score, with the best result corresponding to the highest score.

SECONDARY OUTCOMES:
Active Station Score | The assessment will be conducted at the end of each academic semester, specifically in the 15th week after the beginning of the semester, in accordance with the institution's academic calendar.
  After one minute of reading a simulated clinical case, the student will perform a periapical radiograph using an artificial dental skull model. During this activity, the student is expected to correctly apply biosafety and radioprotection principles, as well as the procedures for radiograph acquisition and processing. At this station, the student will be assessed using a structured checklist with predefined criteria, receiving a score ranging from 0 to 100 points, with 100 representing the highest performance. This station has a total duration of six minutes.
First Passive Station Score | The assessment will be conducted at the end of each academic semester, specifically in the 15th week after the beginning of the semester, in accordance with the institution's academic calendar.
  After one minute of reading a simulated case, the student will interpret a periapical radiograph. They must describe the radiographic technique used, identify the side imaged (right or left; maxillary or mandibular arch), indicate the numerical notation of the teeth shown, and name the visible anatomical structures. At this station, the student will be assessed using a structured checklist with predefined criteria, receiving a score ranging from 0 to 100 points, with 100 representing the highest performance. This station has a total duration of six minutes.
Second Passive Station Score | The assessment will be conducted at the end of each academic semester, specifically in the 15th week after the beginning of the semester, in accordance with the institution's academic calendar.
  After one minute of reading a clinical case, the student will interpret a periapical radiograph, describing the technique used, the side imaged, the numerical notation of the teeth present, and identifying the anatomical structures shown. At this station, the student will be assessed using a structured checklist with predefined criteria, receiving a score ranging from 0 to 100 points, with 100 representing the highest performance. This station has a total duration of six minutes.
Third Passive Station Score | The assessment will be conducted at the end of each academic semester, specifically in the 15th week after the beginning of the semester, in accordance with the institution's academic calendar.
  After one minute of reading a clinical case, the student will interpret the periapical radiograph, describing the radiographic technique, the side imaged, the dental notation, and anatomical structures. Additionally, they must classify the bone defect shown in the image and comment on the etiological factor related to the observed periodontal condition. At this station, the student will be assessed using a structured checklist with predefined criteria, receiving a score ranging from 0 to 100 points, with 100 representing the highest performance. This station has a total duration of six minutes.
Fourth Passive Station Score | The assessment will be conducted at the end of each academic semester, specifically in the 15th week after the beginning of the semester, in accordance with the institution's academic calendar.
  After one minute of reading, the student will interpret the periapical radiograph, describing the technique used, the side imaged, dental notation, and anatomical structures. Additionally, they must assess, based on the image, the need for tooth extraction and prepare a complete radiographic report. At this station, the student will be assessed using a structured checklist with predefined criteria, receiving a score ranging from 0 to 100 points, with 100 representing the highest performance. This station has a total duration of six minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Juiz de Fora, Juiz de Fora, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stellefson M, Paige SR, Chaney BH, Chaney JD. Evolving Role of Social Media in Health Promotion: Updated Responsibilities for Health Education Specialists. Int J Environ Res Public Health. 2020 Feb 12;17(4):1153. doi: 10.3390/ijerph17041153. PMID 32059561
- [Background] Soltanimehr E, Bahrampour E, Imani MM, Rahimi F, Almasi B, Moattari M. Effect of virtual versus traditional education on theoretical knowledge and reporting skills of dental students in radiographic interpretation of bony lesions of the jaw. BMC Med Educ. 2019 Jun 25;19(1):233. doi: 10.1186/s12909-019-1649-0. PMID 31238927
- [Background] Rajeh MT, Sembawa SN, Nassar AA, Al Hebshi SA, Aboalshamat KT, Badri MK. Social media as a learning tool: Dental students' perspectives. J Dent Educ. 2021 Apr;85(4):513-520. doi: 10.1002/jdd.12478. Epub 2020 Nov 20. PMID 33219515
- [Background] Neiva GF, Hasslen JA, Bompolaki D, Pugach-Gordon M, Wright W, Kumar SS. Social media in dental education: The need for institutional policies and content regulation. J Dent Educ. 2023 Oct;87(10):1476-1480. doi: 10.1002/jdd.13310. Epub 2023 Jul 7. No abstract available. PMID 37419870
- [Background] McAndrew M, Johnston AE. The role of social media in dental education. J Dent Educ. 2012 Nov;76(11):1474-81. PMID 23144483
- [Background] Latif MZ, Hussain I, Saeed R, Qureshi MA, Maqsood U. Use of Smart Phones and Social Media in Medical Education: Trends, Advantages, Challenges and Barriers. Acta Inform Med. 2019 Jun;27(2):133-138. doi: 10.5455/aim.2019.27.133-138. PMID 31452573
- [Background] Kumar V, Gadbury-Amyot CC. Predoctoral Curricular Revision for Dental Radiographic Interpretation Competence Based on OSCE Results. J Dent Educ. 2019 Oct;83(10):1233-1239. doi: 10.21815/JDE.019.112. Epub 2019 Jun 10. PMID 31182621
- [Background] Kenny P, Johnson IG. Social media use, attitudes, behaviours and perceptions of online professionalism amongst dental students. Br Dent J. 2016 Nov 18;221(10):651-655. doi: 10.1038/sj.bdj.2016.864. PMID 27857111
- [Background] Kalantari M, Zadeh NL, Agahi RH, Navabi N, Hashemipour MA, Nassab AHG. Measurement of the levels anxiety, self-perception of preparation and expectations for success using an objective structured clinical examination, a written examination, and a preclinical preparation test in Kerman dental students. J Educ Health Promot. 2017 May 5;6:28. doi: 10.4103/jehp.jehp_97_15. eCollection 2017. PMID 28584828
- [Background] Harden RM, Stevenson M, Downie WW, Wilson GM. Assessment of clinical competence using objective structured examination. Br Med J. 1975 Feb 22;1(5955):447-51. doi: 10.1136/bmj.1.5955.447. PMID 1115966
- [Background] Graham R, Zubiaurre Bitzer LA, Mensah FM, Anderson OR. Dental student perceptions of the educational value of a comprehensive, multidisciplinary OSCE. J Dent Educ. 2014 May;78(5):694-702. PMID 24789829
- [Background] Dias da Silva MA, Pereira AC, Walmsley AD. Who is providing dental education content via YouTube? Br Dent J. 2019 Mar;226(6):437-440. doi: 10.1038/s41415-019-0046-8. PMID 30903071
- [Background] Chan TM, Dzara K, Dimeo SP, Bhalerao A, Maggio LA. Social media in knowledge translation and education for physicians and trainees: a scoping review. Perspect Med Educ. 2020 Feb;9(1):20-30. doi: 10.1007/s40037-019-00542-7. PMID 31834598
- [Background] Arnett MR, Christensen HL, Nelson BA. A school-wide assessment of social media usage by students in a US dental school. Br Dent J. 2014 Nov;217(9):531-5. doi: 10.1038/sj.bdj.2014.956. PMID 25377826
- [Background] Almomani EY, Qablan AM, Atrooz FY, Almomany AM, Hajjo RM, Almomani HY. The Influence of Coronavirus Diseases 2019 (COVID-19) Pandemic and the Quarantine Practices on University Students' Beliefs About the Online Learning Experience in Jordan. Front Public Health. 2021 Jan 13;8:595874. doi: 10.3389/fpubh.2020.595874. eCollection 2020. PMID 33520916